CLINICAL TRIAL: NCT05078957
Title: Microbiota Footprint and Frailty Phenotype in Virologically Suppressed People Living With HIV
Acronym: FRAMIVIH
Status: Recruiting | Type: Observational
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 21-33
Record Dates: First submitted 2021-09-17; First posted 2021-10-15 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Frail PLWH
  Interventions: Other: Stool sampling; Other: Frailty phenotype; Other: Blood plasma collection
- Pre frail PLWH
  Interventions: Other: Stool sampling; Other: Frailty phenotype; Other: Blood plasma collection
- No frail PLWH
  Interventions: Other: Stool sampling; Other: Frailty phenotype; Other: Blood plasma collection

INTERVENTIONS:
Other: Stool sampling — Stool samples will be collected from participants at baseline and annually during 5 years
Other: Frailty phenotype — According to Fried frailty phenotype based on the assessment of 5 criteria: shrinking (unintentional weight loss), weakness (grip strength), poor endurance (exhaustion), slowness (walking speed) and physical activity. Frail phenotype is defined as the presence of at least 3 criteria of the above mentioned and Pre-frail phenotype as the presence of 1 or 2 criteria.
Other: Blood plasma collection — Blood plasma collection to measure persistent inflammation and immune activation

SUMMARY:
Analysis of gut microbiota becomes more and more accessible in recent years. Experimental data in both animal and human studies have demonstrated that imbalance of the gut microbiota which is called symbiosis may participate in an accelerated procedure of ageing as well as the expression of frailty phenotype. People living with HIV (PLHIV) present markers of phenotypic frailty on average 10 years before uninfected people.

In this population structural and functional modifications of GALT (Gut Associated Lymphoid Tissue) are observed early after HIV infection and persist despite virological suppression on ART (AntiRetroviral Treatment). These GALT modifications are associated with microbial translocation that is also correlated with immune activation and dysbiosis.

The objective of study is to explore gut microbiota of PLWH over 5 years, as well as to study associations of its longitudinal evolution with frailty markers and burden of comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Individuals infected with HIV in the stable phase of their disease (absence of disease outbreak and absence of therapeutic modification within 3 months before inclusion),
* Subject with ongoing HIV follow-up on an outpatient basis (outpatient or day hospital consultation) in the participating center, and having virological suppression at the threshold of 50 copies / mL for at least 5 years (tolerance of blips < 200 copies / mL during this period)
* Aged ≥ 55 at baseline
* CD4 + T cell nadir> 200 / mm3
* Giving free and informed written consent
* Being affiliated with or benefiting from a social security scheme.

Exclusion Criteria:

* Persons treated with antibiotics, probiotics, prebiotics or any other treatment that may disrupt the gut microbiota within two months before stool sampling.
* Subject not followed regularly in the participating center,
* Subject only coming for full hospitalization
* Subject in the primary infection phase of less than 1 year

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People Living with HIV (PLWH)
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Variation of the Shannon index between 0 and 5 years in different groups of PLWH | Five years

SECONDARY OUTCOMES:
Variation of the Shannon index between 0 and 3 years in different groups of PLWH (frail, pre frail, not frail) | Three years
Assaying inflammation markers(CRP, IL-6, sCD14, sCD163, TNFa, IP10, I-FABP, LBP, D-dimers, K/T ratio) annually and for 5 years in different groups of PLWH | Five years
Correlation between the Shannon index and the number of comorbidities associated with 0, 3 and 5 years in the different groups of PLWH | Five years

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Européen Marseille, Marseille, France